CLINICAL TRIAL: NCT03771261
Title: Balanced (Egg) Protein During Obesity Reduction: Differential Responses of Insulin Resistance by Race
Acronym: EGGSPDITe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00089075
Record Dates: First submitted 2018-11-21; First posted 2018-12-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2022-01

CONDITIONS: Pre Diabetes; Obesity
Keywords: Egg; Protein; Aging; Health Disparities; Weight Loss
MeSH Terms: conditions — Glucose Intolerance; Obesity; Weight Loss | interventions — Egg Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WL-Control (Placebo Comparator): Weight loss intervention (WL-Control; n = 20): Subjects follow a calorie-reduction diet for a weight loss of ≥10%, protein~0.8g/g/d.
  Interventions: Behavioral: Weight Loss
- WL-Protein (Active Comparator): High-protein weight loss intervention (WL-Protein; n = 20): Subjects follow a calorie-reduction diet for a weight loss of ≥10%, with a high proportion of high quality protein at each meal. Intakes of > 30g of protein will be achieved three times a day by subjects in this group, with all or predominantly all from animal sources (high quality) and 60-70% of animal protein from eggs or egg protein powder that will be provided to WL-Protein participants.
  Interventions: Behavioral: Weight Loss; Dietary Supplement: Egg Protein

INTERVENTIONS:
Behavioral: Weight Loss — Participants will be prescribed hypo-caloric diet by a registered dietitian and attend weekly social support/nutrition education meetings.
Dietary Supplement: Egg Protein — Participants will be provided pre-packaged hard-boiled eggs (3/day, medium) and egg white protein powder.
  Arms: WL-Protein

SUMMARY:
The purpose of the trial is to assess the effects of combining regular, generous intakes of high quality protein (with substantial amounts provided from whole eggs and egg whites) with calorie restriction on insulin resistance and weight loss (along with function, body composition, racial disparities, and a number of secondary outcomes) in black and white older adults with prediabetes who are participating in a 4-month intervention. The investigators will compare these effects to the same outcomes with a control group consuming a traditional control regimen of calorie restriction over the same duration.

DETAILED DESCRIPTION:
Older (>60 yrs) men and women (50% African American, 50% white) who are obese (BMI >30 kg/m2) and have pre-diabetes will be randomly assigned (1:1 ratio; couples randomized together) to one to two treatment groups: 1) Weight loss intervention (WL-Control; n = 20): subjects follow a calorie-reduction diet for a weight loss of ≥10%, protein~0.8g/g/d; and 2) High protein weight loss intervention (WL-Protein; n = 20): subjects follow a calorie-reduction diet for a weight loss of ≥10%, with a high proportion of high quality protein (> 30g protein, 3/day, 60-70% egg protein). Primary (insulin resistance/sensitivity, weight loss) and secondary outcomes (physical function, body composition, diet adherence, cognitive function, readiness to change) will be measured at 0 and 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Identifies as Caucasian/white or African-American/black
* Obese body weight (>30 kg/m2)
* Able to speak and understand spoken and written English
* Elevated fasting plasma glucose (≥95 and <126 mg/dL)
* Age-normal Kidney function (≥ 45 mL/min/1.73 m2)

Exclusion Criteria:

* Body weight > 224 kg (limit of the BodPod)
* Treated or untreated diabetes (prior diagnosis, treatment, or fasting blood glucose ≥126 mg/dL)
* Presence of unstable, acutely symptomatic, or life-limiting illness
* Positive screen for dementia using Mini-Cog evaluation tool
* Neurological conditions causing functional or cognitive impairments
* History of significant weight instability (defined as > 10 pounds weight gain or loss over 6 months prior to study participation)
* Allergy or intolerance to egg products
* Unwillingness or inability to be randomized to any one of two intervention groups, submit to all study testing, or continuously participate in a randomly assigned lifestyle intervention program for four months
* Inability to walk independently
* Unable to give consent
* Unable to complete written recording forms including journals of eating and exercise behaviors.
* Current use of the following medications: monoamine oxidase inhibitors, prescription weight loss medications, insulin, metformin or any other hypoglycemic agent
* Primary Care Physician advises against participation
* Smoker
* Unusually or unstable renal function

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Insulin Resistance at 4 months | 0 to 4 months
  Blood glucose and insulin levels in whole blood will be used to compute HOMA-IR (= glucose mg/dL x insulin mg/dL/405)
Change from Baseline Body weight at 4 months | 0 to 4 months
  Weight loss as measured in light clothing on a dedicated scale.

SECONDARY OUTCOMES:
Change from baseline Short Physical Performance Battery at 4 months | 0 to 4 months
  Physical Performance as measured by Short Physical Performance Battery (SPPB)
Change from baseline 6-minute walk (meters) at 4 months | 0 to 4 months
  Distance (meters) walked in 6 minutes
Change from baseline 8-foot up and Go time at 4 months | 0 to 4 months
  Time it takes to get up from a chair walk around a cone and sit back down (8-foot up and go)
Change from baseline 30-second chair stands (number of stands) at 4 months | 0 to 4 months
  the number of chair stands completed in 30 seconds
Change from baseline handgrip strength at 4 months | 0 to 4 months
  the highest weight achieved from 2 attempts using the JAMAR dynamometer
Change from baseline grooved pegboard time at 4 months | 0 to 4 months
  measure of hand dexterity, time it takes to fit pegs into grooved pegboard
Change from baseline fat mass (%) at 4 months | 0 to 4 months
  Body fat mass (%) as measured by Bodpod
Change from baseline fat mass (kgs) at 4 months | 0 to 4 months
  Body fat mass (kg) as measured by Bodpod
Change from baseline lean mass (kgs) at 4 months | 0 to 4 months
  Body lean mass (kg) as measured by Bodpod
Change from baseline lean mass (%) at 4 months | 0 to 4 months
  Body lean mass (%) as measured by Bodpod
Change from baseline minimal waist circumference at 4 months | 0 to 4 months
  Body proportions will be measured at the minimal waist using a Gulick II tape measure with the tape placed directly on the skin (not over the clothing). Measurements will be taken once at each location before completing a second measurement, and an average of the two will be recorded. A third measurement will be taken if the first two measurements are > 0.5 cm.
Change from baseline umbilical waist circumference at 4 months | 0 to 4 months
  Body proportions will be measured at the umbilical waist using a Gulick II tape measure with the tape placed directly on the skin (not over the clothing). Measurements will be taken once at each location before completing a second measurement, and an average of the two will be recorded. A third measurement will be taken if the first two measurements are > 0.5 cm.
Change from baseline hip circumference at 4 months | 0 to 4 months
  Body proportions will be measured at the hip using a Gulick II tape measure with the tape placed directly on the skin (not over the clothing). Measurements will be taken once at each location before completing a second measurement, and an average of the two will be recorded. A third measurement will be taken if the first two measurements are > 0.5 cm.
Change from baseline total calories at 4 months | 0 to 4 months
  Total calories will be measured using 3-day food records (participants record everything they eat and drink for three days)
Change from baseline macronutrient intake at 4 months | 0 to 4 months
  Macronutrient intake will be measured using 3-day food records (participants record everything they eat and drink for three days)
Change from baseline micronutrient intake at 4 months | 0 to 4 months
  Micronutrient intake will be measured using 3-day food records (participants record everything they eat and drink for three days)
Change from baseline Symbol digit modalities test at 4 months | 0 to 4 months
  Symbol Digit Modalities Test measures cognitive impairment
Change from baseline Trail Making Test at 4 months | 0 to 4 months
  Trail Making Test neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.
Change from baseline Hopkins Verbal Learning Test at 4 months | 0 to 4 months
  Hopkins Verbal Learning Test consists of three trials of free-recall of a 12-item, semantically categorized list, followed by yes/no recognition.
Change from baseline Profile of Mood States at 4 months | 0 to 4 months
  Profile of Mood States is a psychological rating scale used to assess transient, distinct mood states that uses a five-point scale ranging from "not at all" to "extremely".
Change from baseline Perceived Stress Scale at 4 months | 0 to 4 months
  Perceived Stress Scale is a a 12-item stress assessment instrument. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Change from Baseline Insulin Sensitivity at 4 months | 0 to 4 months
  insulin sensitivity HOMA-β (= 360 x insulin mg/dL / glucose mg/dL - 63; %).

CONTACTS AND LOCATIONS:
Overall Officials: Connie Bales, RD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porter Starr KN, McDonald SR, Bales CW. Obesity and physical frailty in older adults: a scoping review of lifestyle intervention trials. J Am Med Dir Assoc. 2014 Apr;15(4):240-50. doi: 10.1016/j.jamda.2013.11.008. Epub 2014 Jan 17. PMID 24445063
- [Background] Porter Starr KN, Pieper CF, Orenduff MC, McDonald SR, McClure LB, Zhou R, Payne ME, Bales CW. Improved Function With Enhanced Protein Intake per Meal: A Pilot Study of Weight Reduction in Frail, Obese Older Adults. J Gerontol A Biol Sci Med Sci. 2016 Oct;71(10):1369-75. doi: 10.1093/gerona/glv210. Epub 2016 Jan 18. PMID 26786203
- [Background] Porter Starr KN, McDonald SR, Weidner JA, Bales CW. Challenges in the Management of Geriatric Obesity in High Risk Populations. Nutrients. 2016 May 4;8(5):262. doi: 10.3390/nu8050262. PMID 27153084
- See also: Duke University School of Medicine — https://medschool.duke.edu/
- See also: Egg Nutrition Center — https://www.eggnutritioncenter.org/